CLINICAL TRIAL: NCT02036554
Title: To Evaluate Prevention Effect Of Everolimus and Low-dose Tacrolimus in Comparison With Standard-dose Tacrolimus Therapy With Mycophenolic Acid on the New Onset Diabetes Mellitus After Transplantation in the Renal Allograft Recipients
Brief Title: Evaluate Efficacy Study of Combination Therapy of Everolimus and Low Dose Tacrolimus in Renal Allograft Recipients
Acronym: PROTECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, ChulWoo Yang, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AKR11T
Record Dates: First submitted 2013-12-23; First posted 2014-01-15 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Kidney; Complications, Allograft
MeSH Terms: interventions — Everolimus; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus plus Everolimus (Experimental): Low dose Tacrolimus + Everolimus
  Interventions: Drug: Everolimus; Drug: Tacrolimus
- Tacrolimus plus Mycophenolic acid (Active Comparator): standard dose Tacrolimus + Mycophenolic acid
  Interventions: Drug: Tacrolimus; Drug: Mycophenolic acid

INTERVENTIONS:
Drug: Everolimus — Decrease the level of Tacrolimus and add on Everolimus instead of Mycophenolic acid which is standard treatment.
  Other Names: Certican
  Arms: Tacrolimus plus Everolimus
Drug: Tacrolimus — Decrease the level of Tacrolimus and add on Everolimus instead of Mycophenolic acid which is standard treatment.
  Other Names: Tacroli
Drug: Mycophenolic acid — Decrease the level of Tacrolimus and add on Everolimus instead of Mycophenolic acid which is standard treatment.
  Other Names: Cellcept
  Arms: Tacrolimus plus Mycophenolic acid

SUMMARY:
To evaluate prevention effect of combination therapy of Everolimus and low-dose Tacrolimus in comparison with standard-dose Tacrolimus therapy with Mycophenolic acid on the New Onset Diabetes Mellitus after transplantation in the renal allograft recipients

DETAILED DESCRIPTION:
An open-label, randomized, multi-center, comparative parallel study to evaluate prevention effect of combination therapy of Everolimus and low-dose Tacrolimus in comparison with standard-dose Tacrolimus therapy with Mycophenolic acid on the New Onset Diabetes Mellitus after transplantation in the renal allograft recipients: PROTECT study

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 year old
2. At least 3 months after kidney transplantation
3. Subject who is using Tacrolimus ± purine synthesis inhibitor + steroid without change within the past 3 months (except the dosage)
4. MDRD eGFR ≥ 50 mL/min or serum creatinine < 2.0mg/dL within the past 3 months in the 6months after kidney transplantation
5. Rate of change of serum creatinine < +30% within the past 3 months in the 6months after kidney transplantation (if serum creatinine decreased, without rate of change is inclusion possible. if serum creatinine result was normal,regardless of the rate of change is able to register.)
6. Urine protein/creatinine ratio < 1g/g Cr (spot urine) Subject who is not applicable to the diagnostic criteria NODAT on
7. the baseline in the 6months after kidney transplantation
8. Subjects who agree with written informed consent

Exclusion Criteria:

1. Subjects who received combined non-renal transplantation
2. Subject who received re-transplantation
3. ABO blood group incompatible(when anti-ABO Antibody titer <1:128 is inclusion possible.)
4. Sensitized patients before transplantation

   * Pretransplant or peak PRA titer > 50%
   * Pretransplant T cell cytotoxicity crossmatch (+)
5. HLA-identical living related donor
6. Subject who has diabetes mellitus / NODAT before transplantation
7. Subject who has suffered acute rejection episode within the past 3 months in the 6months after kidney transplantation
8. Subject with hypersensitivity to everolimus
9. Subject who should continue nephrotoxic drug until enrollment (Aminoglycoside, amphotericin B, cisplatin)
10. Subject with GI disorder that might interfere with the ability to absorb oral medication. (eg, gastrectomy or insufficiently treated diabetic gastroenteropathy)
11. Subjects with active peptic ulcer
12. HIV, HBsAg, or HCV Ab tests (+)
13. Abnormal liver function test (AST or ALT or total bilirubin> upper normal limit x3)
14. ANC <1.5*109/L or WBC <2.5*109/L or platelet <75*109/L
15. Treatment with an investigational drug within 30 days preceding the first dose of trial medication
16. Women who are either pregnant, lactating, planning to become pregnant in the next 12 months.
17. Subjects with history of cancer(except successfully treated), localized nonmelanocytic skin cancer, PTLD(Post-transplant lymphoproliferative disorder)
18. Subjects with clinically significant infections within the past 4 weeks in the 6months after kidney transplantation
19. Subjects who took major surgery within the past 4 weeks in the 6months after kidney transplantation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Development of NODAT (Fasting glucose ≥ 126 mg/dL, Random glucose ≥ 200 mg/dL) at 12 months | 0 to 12 month
  To evaluate prevention effect of combination therapy of Everolimus and low-dose Tacrolimus in comparison with standard-dose Tacrolimus therapy with Mycophenolic acid on the New Onset Diabetes Mellitus after transplantation at 12 months after date of randomization.

SECONDARY OUTCOMES:
Insulin resistance by HOMA-IR | 0 to 12 months
  Change from Baseline(V2) in Insulin resistance by HOMA-IR at 12months(V6)
Insulin secretion by HOMA-beta | 0 to 12 months
  Change from Baseline(V2) in insulin secretion by HOMA-beta at 12 months(V6)
OGTT (Fasting and PP2hr) | 0 to 12 months
  Change from baseline in OGTT (Fasting and PP2hr) at 12 months(V6)
Needs for anti-diabetic medication or insulin | at Baseline(V2)
  Needs for anti-diabetic medication or insulin at Baseline(V2)
Needs for anti-diabetic medication or insulin at 3 month(V3) | at 3 month(V3)
  Needs for anti-diabetic medication or insulin at 3 month(V3)
Needs for anti-diabetic medication or insulin at 6 month(V4) | at 6 month(V4)
  Needs for anti-diabetic medication or insulin at 6 month(V4)
Needs for anti-diabetic medication or insulin at 9 month(V5) | at 9 month(V5)
  Needs for anti-diabetic medication or insulin at 9 month(V5)
Needs for anti-diabetic medication or insulin at 12 month(V6) | at 12 month(V6)
  Needs for anti-diabetic medication or insulin at 12 month(V6)
Creatinine clearance (MDRD eGFR) at Baseline(V2) | at Baseline(V2)
  Creatinine clearance (MDRD eGFR) at Baseline(V2)
Creatinine clearance (MDRD eGFR) at 3 month(V3) | at 3 month(V3)
  Creatinine clearance (MDRD eGFR) at 3 month(V3)
Creatinine clearance (MDRD eGFR) at 6 month(V4) | at 6 month(V4)
  Creatinine clearance (MDRD eGFR) at 6 month(V4)
Creatinine clearance (MDRD eGFR) at 9 month(V5) | at 9 month(V5)
  Creatinine clearance (MDRD eGFR) at 9 month(V5)
Creatinine clearance (MDRD eGFR) at 12 month(V6) | at 12 month(V6)
  Creatinine clearance (MDRD eGFR) at 12 month(V6)
12 month graft survival | at 12 months(V6)
  After date of randomization, evaluate graft survival rate at 12 months(V6)
12 month patient survival rate | at 12 months(V6)
  After date of randomization, evaluate patient survival rate at 12 months(V6)
Change from baseline in Microalbuminuria(MAU) at 12 months | at 12 months(V6)
  Change from baseline in Microalbuminuria(MAU) at 12 months
Proportion of patients with significant proteinuria greater than 1g/gCr at Baseline(V2) | at Baseline(V2)
  Proportion of patients with significant proteinuria greater than 1g/gCr at Baseline(V2)
Proportion of patients with significant proteinuria greater than 1g/gCr at 3 month(V3) | at 3 month(V3)
  Proportion of patients with significant proteinuria greater than 1g/gCr at 3 month(V3)
Proportion of patients with significant proteinuria greater than 1g/gCr at 6 month(V4) | at 6 month(V4)
  Proportion of patients with significant proteinuria greater than 1g/gCr at 6 month(V4)
Proportion of patients with significant proteinuria greater than 1g/gCr at 9 month(V5) | at 9 month(V5)
  Proportion of patients with significant proteinuria greater than 1g/gCr at 9 month(V5)
Proportion of patients with significant proteinuria greater than 1g/gCr at 12 month(V6) | at 12 month(V6)
  Proportion of patients with significant proteinuria greater than 1g/gCr at 12 month(V6)
Number of episode of biopsy proven acute rejection (BPAR) | at 12 month(V6)
  Cumulative incidence rate of Biopsy Proven Acute Rejection(BPAR) at 12months(V6) after date of randomization.
Number of hospitalization of any cause (except admission for protocol biopsy) at Baseline(V2) | at Baseline(V2)
  Number of hospitalization of any cause (except admission for protocol biopsy) at Baseline(V2)
Number of hospitalization of any cause (except admission for protocol biopsy) at 3 month(V3) | at 3 month(V3)
  Number of hospitalization of any cause (except admission for protocol biopsy) at 3 month(V3)
Number of hospitalization of any cause (except admission for protocol biopsy) at 6 month(V4) | at 6 month(V4)
  Number of hospitalization of any cause (except admission for protocol biopsy) at 6 month(V4)
Number of hospitalization of any cause (except admission for protocol biopsy) at 9 month(V5) | at 9 month(V5)
  Number of hospitalization of any cause (except admission for protocol biopsy) at 9 month(V5)
Number of hospitalization of any cause (except admission for protocol biopsy) at 12 month(V6) | at 12 month(V6)
  Number of hospitalization of any cause (except admission for protocol biopsy) at 12 month(V6)
Number of opportunistic infections (BKVN) at Baseline(V2) | at Baseline(V2)
  Number of opportunistic infections (BKVN) at Baseline(V2)
Number of opportunistic infections (BKVN) at 12month(V6) | at 12 month(V6)
  Number of opportunistic infections (BKVN) at 12month(V6)
Prevalence of NODAT at Baseline(V2) | at Baseline(V2)
  Prevalence of NODAT at Baseline(V2)
Prevalence of NODAT at 3 month(V3) | at 3 month(V3)
  Prevalence of NODAT at 3 month(V3)
Prevalence of NODAT at 6 month(V4) | at 6 month(V4)
  Prevalence of NODAT at 6 month(V4)
Prevalence of NODAT at 9 month (V5) | at 9 month (V5)
  Prevalence of NODAT at 9 month (V5)
Prevalence of NODAT at 12 month(V6) | at 12 month(V6)
  Prevalence of NODAT at 12 month(V6)

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Yang, MD, Principal Investigator — St Mary's Hospital, London
Locations (1):
- division of nephrology;Seoul St Mary's Hospital, Seoul, South Korea